CLINICAL TRIAL: NCT04106648
Title: Effect of Significant Ischemic Mitral Regurgitation on the Outcome of ST Segment Elevation Myocardial Infarction Patients Treated With Primary Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Usama Amin Kostandy, Principal investigator, Assiut University
Other Study IDs: Ischemic mitral regurgitation
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Ischemic Mitral Regurgitation
Keywords: Ischemic Mitral Regurgitation; primary percutaneous coronary intervention; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to correlate the effect of ischemic mitral regurgitation on the outcome of STEMI patients treated with successful primary PCI using clinical data and echocardiography on presentation and during short term follow up after 3 months

DETAILED DESCRIPTION:
* IMR is defined as mitral regurgitation (MR) caused by chronic changes of LV structure and function due to ischemic heart disease. It is not a valve disease but represents the valvular consequences of increased tethering forces and reduced closing forces. It is reported in approximately one-fifth of patients following acute myocardial infarction (MI) and one-half of those with congestive heart failure. IMR is a frequent complication of coronary artery disease and it worsens the prognosis.
* It is important to distinguish between primary MR due to organic disease of one or more components of the mitral valve apparatus and secondary MR which is not a valve disease, but represents LV disease. Secondary MR is defined as functional MR, due to LV remodeling by cardiomyopathy or coronary artery disease. In the latter clinical setting, secondary functional MR is called IMR. There are some limitations in this definition of functional IMR. Recent studies have revealed evidence of structural changes in the mitral leaflets in response to tethering on them by LV pathological remodeling. The leaflet adaptation includes enlargement and increased stiffness.
* Aim of the work :

To correlate the effect of ischemic mitral regurgitation on the outcome of STEMI patients treated with successful primary PCI using clinical data and echocardiography on presentation and during short term follow up after 3 months

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with first presentation
2. Subjects with Acute STEMI
3. Subjects undergoing Primary PCI with Successful reperfusion
4. Subjects with significant IMR Grade (III/IV) to (IV/IV)
5. Subjects with acute STEMI with no or non-significant MR undergoing Primary PCI undergoing primary PCI with successful reperfusion (as control)

Exclusion Criteria:

1. Rheumatic mitral regurge
2. Valvular mitral regurge
3. IMR Grade (II/IV)
4. Cardiomyopathies
5. Associated other valvular heart diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with STEMI undergoing PPCI
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
effect of ischemic mitral regurgitation on the outcome of STEMI patients treated with successful primary PCI | 3 months
  clinical data and echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Fady Usama Kostandy, Msc, Principal Investigator — Assiut University; Hatem Abd El Rahman, Professor, Study Director — Assiut University; Magdy Ibrahim Eldesowky, Lecturer, Study Director — Assiut University

REFERENCES:
- Available data/document: Pubmed — http://www.ncbi.nlm.nih.gov/pubmed/